CLINICAL TRIAL: NCT02250066
Title: Effect of Diet Therapy on Prevention of Type 2 Diabetes Mellitus Among 322 Adults Over 20 Years With Abnormal Glucose Metabolism
Brief Title: Prevention of Type 2 Diabetes Mellitus by Changes in Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilam University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Assistant Professor, MD, Ph.D of Nutrition, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IlamUMS
Record Dates: First submitted 2014-09-17; First posted 2014-09-26 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study group 1 (Other): Received high monounsaturated fat diet
  Interventions: Other: Diet
- Study group 2 (Other): Received high carbohydrate diet
  Interventions: Other: Diet
- Control Group (No Intervention): Control group was encouraged to follow the Food Guide Pyramid

INTERVENTIONS:
Other: Diet — Study group 1 received high monounsaturated fat diet Study group2 received high carbohydrate diet Control group was encouraged to follow the Food Guide Pyramid
  Arms: Study group 1; Study group 2

SUMMARY:
investigators evaluated the efficacy of two types of diet with different macronutrients, on prevention or delaying the onset of type 2 diabetes in subjects with either impaired fasting glucose (IFG) or impaired glucose tolerance (IGT). 322 subjects with prediabetes were randomly assigned to high monounsaturated fat diet (n=107), high carbohydrate diet (n=106) or control group (n=109) and followed for 2 years. For calculating daily energy requirement in subjects with BMI≥25 kg/m2 the weight was adjusted with the use of 110 percent of the ideal body weight with no attempt for losing body weight. Control group were encouraged to follow the Food Guide Pyramid and reduce their fat intake to less than 30% of energy consumed and saturated fat to less than 10 percent of total energy. The primary outcome variable was incidence of type 2 diabetes mellitus, diagnosed by the latest American Diabetic Association criteria.

DETAILED DESCRIPTION:
322 participants were randomized and stratified into a control group and two study groups according to sex, age, body mass index (BMI), IFG and IGT or both. Baseline assessments were anthropometric measurements, food diary and laboratory exams. Anthropometric measurements were repeated annually. Blood sample tests measured fasting blood glucose, glucose two hours after ingestion of 75 g glucose, high density lipoprotein (HDL), low density lipoprotein (LDL) and triglyceride (TG), which were analyzed in the laboratory of the only university hospital in the city. The same assessments were repeated annually (at 12 and 24 months) in all groups. Daily energy requirement was calculated by multiplying 30-35 Kcal per Kg body weight for each participant. For patients with BMI ≥25 kg/m2, the weight was adjusted with use of 110 percent of the ideal body weight. Diet in HCD group was 15% from protein, 30% from fat (10% MUFA, 10% PUFA, 10% SFA) and 55% from carbohydrate. Diet in HMD group was 15% from protein, 45% from fat (25% MUFA, 10% PUFA, 10% SFA) and 40% from carbohydrate. Source of MUFA in this group was olive oil. In the intervention groups diet regimen was written for each participant by a registered dietitian. Group three or the control group was encouraged to follow the Food Guide Pyramid and reduce their fat intake to less than 30 percent of energy consumption and saturated fat to less than 10 percent of total energy.

ELIGIBILITY:
Inclusion Criteria: Adults over 20 years Exclusion Criteria: Diet therapy; severe physical activity; accompanying diseases such as cancer which reduce their life expectancy; receiving thiazide diuretics; receiving systemic ß blockers; receiving glucocorticoids; receiving nicotinic acid; receiving weight lowering drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Diabetes in 322 Subjects with Prediabetes | Up to 24 months

IPD SHARING:
Plan to Share IPD: No